CLINICAL TRIAL: NCT04422405
Title: Functional Changes in the Stomach and Esophagus After One Anastomosis Gastric Bypass- OAGB- BiFlux Trial
Brief Title: Functional Changes in the Stomach and Esophagus After One Anastomosis Gastric Bypass- OAGB
Acronym: BiFLux
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Marko Kraljevic, MD, Principal Investigator, Spital Limmattal Schlieren
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLS-003
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Morbid; GERD; Ulcer, Gastric
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux; Stomach Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing OAGB (Experimental)
  Interventions: Procedure: One Anastomosis Gastric Bypass (OAGB)

INTERVENTIONS:
Procedure: One Anastomosis Gastric Bypass (OAGB) — The procedure is performed laparoscopically. The "GIA" stapler divides the stomach at the junction of the body and antrum. An Ewald tube, roughly the diameter of the esophagus, is passed by the anesthetist and held against the lesser curvature. The division of the stomach against the tube is completed, with 5- 6 lines of staples. The division of the stomach is parallel to the lesser curvature and up to the angle of His. A point is selected on the small bowel about 200 cm distal to the ligament of Treitz. The jejunal loop is brought up antecolic, and the Endo-GIA stapler is used to perform the anastomosis between the stomach and the small bowel at this point. The distal end of the gastric tube is anastomosed to the side of the small bowel.
  Other Names: Mini-Gastric Bypass

SUMMARY:
Evaluation of the functional changes in the stomach and esophagus of patients undergoing One Anastomosis Gastric Bypass (OAGB)

ELIGIBILITY:
Inclusion Criteria:

* BMI> 35 kg/m2
* 2 years of controlled conservative obesity treatment without weight reduction
* patients should give their consent to participate in the study

Exclusion Criteria:

* Less than 2 years of conservative obesity treatment
* cancer
* cirrhosis Child-Pough score A
* Crohn's disease
* serious psychiatric disorder, which led to in-hospital treatment in psychiatric clinic in the past two years
* drug consumption
* non-compliance
* hiatal hernia > 4cm
* gastric pouch < 10cm
* Barett esophagus
* erosive esophagitis Grade C or D according to the Los Angeles Classification
* endoscopically proven gastric stricture
* acid exposition time > 6% (Lyon criteria)
* reflux episodes> 80 /24 hours (Lyon criteria)
* insufficient low esophageal sphincter according to manometry findings
* pathological findings in the impedance pH-metry (acid and non-acid reflux)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2035-05-28 (Estimated); Study Completion 2035-05-28 (Estimated)

PRIMARY OUTCOMES:
Marginal ulcer rates | 2 years post surgery
Marginal ulcer rates | 5 years post surgery
Assessment of age as risk factor for marginal ulcer development | 2 years post surgery
  Age of participants will be measured in years.
Assessment of age as risk factor for marginal ulcer development | 5 years post surgery
  Age of participants will be measured in years
Assessment of gender as risk factor for marginal ulcer development | 2 years post surgery
  The association between gender of participants (male/female) and incidence of marginal ulcers will be assessed.
Assessment of gender as risk factor for marginal ulcer development | 5 years post surgery
  The association between gender of participants (male/female) and incidende of marginal ulcers will be assessed.
Assessment of tobacco use as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the number of participants who are smokers correlates with the incidence of marginal ulcers.
Assessment of tobacco use as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the number of participants who are smokers correlates with the incidence of marginal ulcers.
Assessment of alcohol use as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the number of participants who report alcohol use correlates with the incidence of marginal ulcers.
Assessment of alcohol use as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the the number of participants who report alcohol use correlates with the incidence of marginal ulcers.
Assessment of nonsteroidal antiinflammatory drug (NSAID) use as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the number of participants who report NSAID use correlates with the incidence of marginal ulcers.
Assessment of nonsteroidal antiinflammatory drug (NSAID) use as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the number of participants who report NSAID use correlates with the incidence of marginal ulcers.
Assessment of immunosuppressive medication usage as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the number of participants who report immunosuppressive medication usage correlates with the incidence of marginal ulcers.
Assessment of immunosuppressive medication usage as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the number of participants who report immunosuppressive medication usage correlates with the incidence of marginal ulcers.
Assessment of Helicobacter pylori as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the incidence of Helicobacter pylori proven by biopsy correlates with the incidence of marginal ulcers.
Assessment of Helicobacter pylori as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the incidence of Helicobacter pylori proven by biopsy correlates with the incidence of marginal ulcer.
Assessment of gastroesophageal reflux disease (GERD) as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the incidence of GERD correlates with the incidence of marginal ulcers.
Assessment of gastroesophageal reflux disease (GERD) as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the incidence of GERD correlates with the incidence of marginal ulcers.
Assessment of diabetes mellitus as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the incidence of diabetes mellitus correlates with the incidence of marginal ulcers.
Assessment of diabetes mellitus as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the incidence of diabetes mellitus correlates with the incidence of marginal ulcers.
Assessment of dyslipidemia as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the incidence of dyslipidemia among the participants correlates with the incidence of marginal ulcers.
Assessment of dyslipidemia as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the incidence of dyslipidemia among the participants correlates with the incidence of marginal ulcers.
Assessment of coronary artery disease (CAD) as risk factor for marginal ulcer development | 2 years post surgery
  It will be assessed if the incidence of CAD among the participants correlates with the incidence of marginal ulcers.
Assessment of coronary artery disease (CAD) as risk factor for marginal ulcer development | 5 years post surgery
  It will be assessed if the incidence of CAD among the participants correlates with the incidence of marginal ulcers.

SECONDARY OUTCOMES:
Total weight loss % (TWL) | 2 years post surgery
Total weight loss % (TWL) | 5 years post surgery
Excess weight loss % (EWL) | 2 years post surgery
Excess weight loss % (EWL) | 5 years post surgery
Total BMI loss (TBL) | 2 years post surgery
Total BMI loss (TBL) | 5 years post surgery
Excess BMI loss (EBL) | 2 years post surgery
Excess BMI loss (EBL) | 5 years post surgery
Late morbidity (>30 days) | 30 days post surgery
  Number of surgical complications according to Dindo-Clavien classification
Late morbidity (>30 days) | 5 years
  Number of surgical complications according to Dindo-Clavien classification
Incidence of gastroesopagheal reflux disease (GERD) | 2 years post surgery
  based on upper gastrointestinal endoscopy findings and classified according to the Los Angeles Classification
Incidence of gastroesopagheal reflux disease (GERD) | 5 years post surgery
  based on upper gastrointestinal endoscopy findings and classified according to the Los Angeles Classification
Incidence of Barrett's esophagus | 2 years post surgery
  based on biopsy findings
Incidence of Barrett's esophagus | 5 years post surgery
  based on biopsy findings
Changes of esophageal motor function | 2 years post surgery
  The esophageal motor function will be measured in mmHg via high-resolution manometry.
Changes of esophageal motor function | 5 years post surgery
  The esophageal motor function will be measured in mmHg via high-resolution manometry.
Esophageal acid or bolus exposure | 2 years post surgery
  Measured with impedance-pH Monitoring. Acid exposure (%) is defined as the total time the pH is < 4 divided by the time monitored. Bolus exposure (%) is defined as being analogous to acid exposure by adding the duration of all four reflux subcategories defined by the impedance, and dividing this value by the time monitored.
Esophageal acid or bolus exposure | 5 years post surgery
  Measured with impedance-pH Monitoring. Acid exposure (%) is defined as the total time the pH is < 4 divided by the time monitored. Bolus exposure (%) is defined as being analogous to acid exposure by adding the duration of all four reflux subcategories defined by the impedance, and dividing this value by the time monitored.
Number of acid or alcaline reflux events | 2 years post surgery
  Measured with impedance-pH Monitoring.
Number of acid or alcaline reflux events | 5 years post surgery
  Measured with impedance-pH Monitoring.
Gastrointestinal quality of life (QoL): GIQLI | 2 years post surgery
  The gastrointestinal (QoL) will be measured using the Gastrointestinal Quality of Life Index (GIQLI). The GIQLI is a validated tool to assess health- related quality of life of patients with gastrointestinal disease or patients who undergo gastrointestinal operations. Its scale is 0-128. Higher values indicate a better quality of life outcome.
Gastrointestinal quality of life (QoL): GIQLI | 5 years post surgery
  The gastrointestinal (QoL) will be measured using the Gastrointestinal Quality of Life Index (GIQLI). The GIQLI is a validated tool to assess health- related quality of life of patients with gastrointestinal disease or patients who undergo gastrointestinal operations. Its scale is 0-128. Higher values indicate a better quality of life outcome.
Obesity- related quality of life (QoL): BAROS | 2 years post surgery
  Obesity- related QoL will be measured with the BAROS (Bariatric Analysis and Reporting Outcome System). BAROS consists of a scoring table that includes three columns with the main areas of interest: weight loss, improvement of medical conditions, and QoL. A maximum of three points is given in each domain to evaluate changes after medical intervention (maximum score is 9 points). Higher scores indicate a better outcome.
Obesity- related quality of life: BAROS | 5 years post surgery
  Obesity- related QoL will be measured with the BAROS (Bariatric Analysis and Reporting Outcome System). BAROS consists of a scoring table that includes three columns with the main areas of interest: weight loss, improvement of medical conditions, and QoL. A maximum of three points is given in each domain to evaluate changes after medical intervention (maximum score is 9 points). Higher scores indicate a better outcome.
Reflux-associated symptoms | 2 years post surgery
  GERD symptoms will be measured with the Gastroesophageal reflux disease questionnaire (GERDQ). GERDQ has a scale between 0 and 18 points. Increasing scores correlate with increasing severity of heartburn symptoms.
Reflux-associated symptoms | 5 years post surgery
  GERD symptoms will be measured with the Gastroesophageal reflux disease questionnaire (GERDQ). GERDQ has a scale between 0 and 18 points. Increasing scores correlate with increasing severity of heartburn symptoms.
Reflux-associated quality of life (QoL): GERD-HRQL | 2 years post surgery
  Reflux- associated QoL will be assessed with the Health-related QoL scale for GERD (GERD-HRQL). The scale has 11 items, which focus on heartburn symptoms, dysphagia, medication effects and the patient's present health condition. Each item is scored from 0 to 5, with a higher score indicating a better QoL.
Reflux-associated quality of life (QoL): GERD-HRQL | 5 years post surgery
  Reflux- associated QoL will be assessed with the Health-related QoL scale for GERD (GERD-HRQL). The scale has 11 items, which focus on heartburn symptoms, dysphagia, medication effects and the patient's present health condition. Each item is scored from 0 to 5, with a higher score indicating a better QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Limmattal Hospital, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No